CLINICAL TRIAL: NCT07100834
Title: Pulsed ElectRic FiEld Versus Cryoballoon to Treat Paroxysmal Atrial Fibrillation (PERFECT-PAF) Randomized Trial
Brief Title: Pulsed ElectRic FiEld Versus Cryoballoon for PAF
Acronym: PERFECT-PAF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Carlo de Asmundis, Department Director, Universitair Ziekenhuis Brussel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC-2023-208
Record Dates: First submitted 2025-07-27; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Atril Fibrillation; Cardiac Arrhythmia; Paroxysmal Atrial Fibrillation (PAF)
Keywords: atrial fibrillation; ablation; pulsed field ablation; cryoablation; cryoballoon; paroxysmal atrial fibrillation
MeSH Terms: conditions — Arrhythmias, Cardiac; Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: This is a singlecenter, prospective, randomized, non-inferiority, parallel-group, investigator-initiated trial with blinded endpoint assessment in which up to 202 paroxysmal AF patients will be randomly assigned to receive cryoballoon (Group Cryo; n=101) or pulsed electric field (PEF)-(Group PFA; n=101) ablation for pulmonary vein isolation (PVI).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulsed Field Ablation (Experimental): The FARAPULSE™ Pulsed Field Ablation System (Boston Scientific, Inc.) is a CE-marked system consisting of the FARASTAR™ Pulsed Field Ablation Generator that is used with the FARAWAVE™ Pulsed Field Ablation Catheter for cardiac tissue ablation
  Interventions: Device: Single-Shot Pulsed Field Ablation (FARAPULSE™ Pulsed Field Ablation System)
- Cryoballoon Ablation (Active Comparator): The Arctic Front Advance PRO, POLARx and Polarx FIT Balloon Catheters are CE-marked cryoablation systems consisting of a cryoballoon device, which is used in conjunction with a CryoConsole, a steerable sheath, and a circular mapping catheter
  Interventions: Device: Single-Shot Cryoballoon Devices (Arctic Front Advance PRO, Medtronic Inc., Minneapolis, MN, USA; POLARx and POLARx FIT Balloon Catheter, Marlborough, MA, USA)

INTERVENTIONS:
Device: Single-Shot Pulsed Field Ablation (FARAPULSE™ Pulsed Field Ablation System) — The FARAPULSE™ Pulsed Field Ablation System (Boston Scientific, Inc.) is a CE-marked system consisting of the FARASTAR™ Pulsed Field Ablation Generator that is used with the FARAWAVE™ Pulsed Field Ablation Catheter for cardiac tissue ablation
  Arms: Pulsed Field Ablation
Device: Single-Shot Cryoballoon Devices (Arctic Front Advance PRO, Medtronic Inc., Minneapolis, MN, USA; POLARx and POLARx FIT Balloon Catheter, Marlborough, MA, USA) — The Arctic Front Advance PRO, POLARx and FIT Balloon Catheters are CE-marked cryoablation systems consisting of a cryoballoon device, which is used in conjunction with a CryoConsole, a steerable sheath, and a circular mapping catheter
  Arms: Cryoballoon Ablation

SUMMARY:
This study has been designed to compare the success rate of two different commercially available ablation technologies, namely PFA and Cryo. Both technologies are standard of care ablation procedures. An ablation is a procedure where a small piece of tissue of the heart, that. causes an irregular heartbeat, is heated or frozen (cryo-ablation) using a special type of catheter.

Once you have signed this consent to take part of the study, you will be randomly assigned to one of the two ablation strategies (PFA versus Cryo). Randomization is a method that helps prevent any possible influence of human choices on clinical results and improve objectivity in research. The day of the procedure you will be undergo AF catheter ablation via either PFA or Cryo based on the results of randomization.

Although both devices that will be used in this study are commercially approved, assessing the incidence of arrhythmia recurrence after ablation during follow-up is considered the investigational portion of the study. "Investigational" means that recurrence data will be collected after the cardiac ablation procedure and compared amongst the two standard of care ablation methods used to treat AF. This study will investigate how well PFA and Cryo work to prevent recurrences of atrial arrhythmias and if there are any differences between the two technologies

DETAILED DESCRIPTION:
AF is the most common sustained arrhythmia, substantially increasing morbidity and mortality, in addition of being a significant burden on healthcare systems worldwide. During the last decades, catheter ablation with radiofrequency (RF) energy has emerged as an alternative non-pharmacological therapy for AF patients who are intolerant to AADs.2 Catheter ablation is currently the most effective rhythm control strategy;3 its rationale lies in the elimination of atrial sites involved in AF initiation/maintenance. Specifically, studies have demonstrated a critical role of pulmonary veins (PVs) as a source of ectopic beats triggering AF paroxysms and that isolation of PVs (PVI) from the left atrium effectively prevents atrial tachyarrhythmia relapse in paroxysmal AF patients. In addition to point-by-point isolation, PVI can also be achieved with single-shot technologies (e.g., cryoballoon, RF balloon, laser balloon), which have been developed aiming at simplifying the procedure and minimizing the influence of operator's experience on procedural safety and success.

Cryoballoon ablation is currently the most widespread single-shot technique for PVI. Its safety and efficacy has been demonstrated to be superior to antiarrhythmic drug treatment4,5 and non-inferior to RF-based point-by-point PVI in randomized and non-randomized trials.

Both RF and cryothermy rely on thermal processes (heating or freezing, respectively) for cardiac tissue death induction. Despite significant technological improvements and a better understanding of the biophysics of thermal ablation, the main shortcoming of these techniques is the lack of tissue selectivity. Achieving contiguous, transmural cardiac lesions may be associated to an increased risk of collateral damage to surrounding tissues (e.g., phrenic nerve, esophagus, blood vessels).

PFA has emerged as a novel ablation technology, which involves the application of ultrarapid (microseconds to nanoseconds), high-amplitude electrical pulses. These pulses generate strong electric fields with an increase in cell membrane permeability and impaired cell homeostasis, which may promote cell death. In this perspective, PFA differs from the above-mentioned thermal energy sources since it does not rely on thermal processes to achieve ablation. Moreover, the treatment protocol can be designed to overcome/limit the risk of collateral tissue damage and improve cardiac lesion durability.

To date, the only PFA device with regulatory approval (CE-mark) is the multielectrode Farawave catheter (FarapulseTM-Boston Scientific Inc., Marlborough, Massachusetts, USA). The safety and efficacy of the system has been tested in two phase 3 studies enrolling paroxysmal and persistent AF patients, which demonstrated remarkable safety and lesion durability results. Similar observations were confirmed in multiple subsequent post-approval registries.

In addition, the safety and efficacy of the pentaspline FarapulseTM PFA catheter has been reported in several registries12,14, as well as a recent randomized study10 comparing this new technology versus traditional energy sources (e.g. radiofrequency and cryothermy). Our group has been actively involved since the earliest stages of the release of the Farapulse technology. We are one of the two sites worldwide to have all three approved PFA technologies. Our center experience with the FarapulseTM technology includes >600 atrial fibrillation procedures. All operators involved in the trial have performed at least 50 PFA cases and are considered opinion leaders in the field and with the technology.

Nonetheless, no data currently exist directly comparing the safety and long-term efficacy of single-shot PFA versus cryoballoon ablation. This study is designed to compare the well-established approach of cryoballoon ablation with the novel PFA-based single-shot Farapulse device for PVI of PAF in a randomized fashion.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of recurrent symptomatic non-valvular paroxysmal AF (PAF);
2. Age 18 through 75 years-old on the day of enrollment;
3. Willing and capable of providing written informed consent;
4. Willing and capable of complying with all pre-, post- and follow-up testing andrequirements.

Exclusion Criteria:

1. AF secondary to electrolyte imbalance, thyroid disease, valvular disease, or reversible or non-cardiac cause;
2. Previous left atrium (LA) ablation or surgery;
3. Previously diagnosed with persistent AF (greater than [>] 7 days in duration);
4. Severe dilatation of the LA (LAD >50 millimeter (mm) antero-posterior diameter in case of transthoracic echocardiography (TTE));
5. Pregnant or lactating (current or anticipated) at the time of catheter ablation;
6. Current enrollment in any other study protocol where testing or results from that study may interfere with the procedure or outcome measurements for this study;
7. Any other conditions such as, mental illness, addictive disease, terminal illness with a life expectancy of less than two years, extensive travel away from the research center that may lead to non-compliance with the protocol procedure or follow up.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2023-09-27 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint | 0-36 months
  the primary efficacy endpoint will be the incidence of any atrial tachyarrhythmia (AF, atrial flutter, atrial tachycardia) lasting >30s during at least 1 year of follow-up. Recurrences occurring within the first 90 days post-ablation (the so-called "blanking period") will not be considered for primary efficacy endpoint measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Domenico G Della Rocca, MD, PhD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (6):
- Universitair Ziekenhuis Brussel, Brussels, Belgium
- Department of Cardiovascular Diseases, University Hospital Center Zagreb, Zagreb, Croatia
- 9. First Department of Cardiology, National and Kapodistrian University of Athens Medical School, Hippokration General Hospital, Athens, Greece
- Italy (2):
  - Maria Cecilia Hospital, Cotignola
  - Ospedale Fatebenefratelli Isola Tiberina-Gemelli Isola, Roma
- Department of Cardiology, Medical University of Lublin, Lublin, Poland

IPD SHARING:
Plan to Share IPD: Undecided